CLINICAL TRIAL: NCT03632889
Title: A Computerized Cognitive Behavioral Therapy (CBTi) Randomized, Controlled, Pilot Trial for Insomnia in Epilepsy
Brief Title: A Computerized CBTi for Insomnia in Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Nancy Foldvary-Schaefer, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-242
Record Dates: First submitted 2018-07-25; First posted 2018-08-16 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Epilepsy; Insomnia
MeSH Terms: conditions — Epilepsy; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): Subjects randomized to the control group will receive a sleep hygiene handout .
- Computerized Group (Other): Subjects randomized to GoToSleep program will receive a sleep hygiene handout and a unique code for home access to the GoToSleep program.
  Interventions: Behavioral: GoToSleep Program

INTERVENTIONS:
Behavioral: GoToSleep Program — For the control group only the sleep hygiene handout will be given in this arm. For the computerized group a sleep hygiene handout along with assess to the GoToSleep online program.
  Arms: Computerized Group

SUMMARY:
This is a pilot study.

The Investigators propose a pilot randomized, parallel-group, controlled trial comparing the GoToSleep program (GTS) and controls on change in Insomnia Severity Index (ISI) from baseline to week 8 in adults with epilepsy and moderate-to-severe insomnia.

Adults with epilepsy and moderate-to-severe insomnia symptoms (ISI ≥15) 17 will be identified using data collected as part of routine clinical care in the adult epilepsy clinic.

All subjects will be provided a consent form describing the study and provided sufficient information to make an informed decision. After a screening visit, subjects meeting study criteria will be randomized to the computerized cognitive behavioral therapy for insomnia (CCBT-i) using the GoTosleep (GTS) or the control group. Both groups will receive a sleep hygiene handout that is standard of care in the treatment of insomnia. All subjects will be contacted by phone every 2 weeks during the intervention to address questions related to sleep hygiene instructions and use of the CCBT-i in the GoTosleep (GTS) group. All subjects will complete a series of sleep related patient reported outcomes including the ISI at baseline 8 weeks post randomization and maintain a diary recording of seizures and sleep periods. Those randomized to CCBT-i will complete a questionnaire at week 8 assessing barriers to CCBT-i.

Subjects randomized to the control group will be offered access to the GoTosleep (GTS) at no charge at the end of the study (week 8).

DETAILED DESCRIPTION:
Growing interest in the relationship between epilepsy and sleep has resulted in a number of investigations demonstrating the high prevalence of sleep disturbances and disorders in people with epilepsy (PWE). PWE frequently report daytime sleepiness, insomnia, and other sleep problems.

Insomnia is among the most common sleep complaint in PWE. The prevalence of moderate-to-severe insomnia using the ISI ranges from 15% to 51%. A recent case-control study found an association between insomnia symptom severity and poorer seizure control. Difficulty maintaining sleep is the most common insomnia presentation followed by difficulty initiating sleep. Both patterns are accompanied by a decrease in total sleep time and an increase in the number of awakenings, arousals and wake time after sleep onset, leading to a state of relative sleep deprivation. Like epilepsy, insomnia disorders are commonly associated with co-morbid depression in the general population, confirmed in a cohort of adults with epilepsy from our own epilepsy center. In turn, treatment of depression has been shown to improve insomnia in the general population. Further, improved seizure control has been observed following treatment of other comorbid sleep disorders such as obstructive sleep apnea and poor sleep hygiene. Innovative sleep treatments for PWE are needed.

To date, there are no studies exploring sleep and seizure outcomes with treatment of insomnia in PWE. Cognitive Behavioral Therapy for Insomnia(CBT-i) is generally the preferred initial treatment for most cases of primary insomnia. CBT-i examines and promotes modifications in thoughts and behaviors that perpetuate insomnia. The validity of CBT-i has been well established and the American College of Physicians has acknowledged CBT-i as the first-line therapy for insomnia with treatment effects that outlast those of sedative-hypnotic medications. Despite its established efficacy, CBT-i is not widely accessible due to the lack of trained clinicians, stigmatization in receiving psychological services, geographical remoteness to trained providers and cost. Treatment typically involves a series of up to 10 visits at weekly or biweekly intervals.

In recent years, CCBT-i programs have been developed that offer web-based treatment. One such program is GoTo sleep (GTS), developed and validated by investigators at the Cleveland Clinic. GTS constitutes 6 weeks of therapy based on the principles and methods of CBT-i presented as a series of daily lessons, learnable skills, and personalized recommendations supported by graphics, animations, audio and video. The program includes the basic elements of CBT-i including sleep hygiene, sleep restriction, stimulus control, cognitive restructuring and relaxation training. The efficacy of CCBT-i has been demonstrated in several randomized controlled trials involving patients with primary insomnia including one using GTS where the program was found to be superior to usual care (sleep hygiene instruction) after 6 weeks of therapy. Further, we recently conducted a pilot study comparing GTS and standard sleep hygiene instruction in Parkinson's disease patients with insomnia and found a greater reduction in ISI scores with CCBT-i (-7.9 vs -3.5; p=0.03).

Given the prevalence of insomnia in epilepsy and the known association between seizure occurrence and sleep impairment, the investigators hypothesize that treatment of insomnia with CCBT-i will improve insomnia symptoms and seizure control in PWE.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Baseline ISI score ≥15
* Stable antiepileptic drug (AED) therapy for >30 days prior to enrollment without planned medication change, surgery or in-patient testing in the coming 90 days
* Able to quantify seizures
* Daily access to computer and internet
* Sufficient computer skills to engage in the on-line program
* Able to speak, read and understand English

Exclusion Criteria:

* Poorly quantified epileptic seizures, psychogenic non-epileptic seizures or other types of spells of undetermined etiology
* Cognitive impairment judged to be significant enough so as to impair one's ability to adhere to study procedures and sleep recommendations
* Major depression with suicidal ideations or presence of active co-morbid conditions that may affect study participation/completion
* Co-morbid sleep disorders that could be contributing to insomnia symptoms such as sleep apnea, restless legs syndrome (RLS) and circadian rhythm disorders
* Use of sedative-hypnotics, benzodiazepines, psychotropics, wake promoting agents and stimulants will be permitted provided the subject has been on a stable dose for at least 1 month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Primary Aim - To compare change in Insomnia Severity Index (ISI) score from baseline to week 8 between Go! to sleep (GTS) and control in people with epilepsy and moderate-to-severe insomnia. | baseline to 8 weeks
  The number of participants with change in Insomnia Severity Index (ISI) score, total range score of 0-28, from baseline to week 8 in people with epilepsy (PWE)and moderate-to-severe insomnia with Go! To sleep (GTS) program compare to the number of participants with change in Insomnia Severity Index (ISI) score from baseline to week 8 in people with epilepsy (PWE) and moderate-to-severe insomnia without Go! To sleep (GTS) program

SECONDARY OUTCOMES:
Secondary Aim 1 - To compare change in sleep quality on the Pittsburgh Sleep Quality Inventory (PSQI) from baseline to week 8 between Go! To sleep (GTS) and controls in people with epilepsy and moderate-to-severe insomnia symptoms. | Baseline to 8 weeks
  The number of participants with change in sleep quality on the Pittsburgh Sleep Quality Inventory (PSQI) score (total score range of 0-21), from baseline to week 8 in people with epilepsy (PWE) and moderate-to-severe insomnia with Go! To sleep (GTS) program compare to the number of participants with change in sleep quality on the Pittsburgh Sleep Quality Inventory (PSQI) score from baseline to week 8 in people with epilepsy (PWE) and moderate-to-severe insomnia without Go! To sleep (GTS) program
Secondary Aim 2 - To compare change in fatigue symptom on the Fatigue Severity Scale (FSS) from baseline to week 8 between Go! To sleep (GTS) and controls in people with epilepsy and moderate-to-severe insomnia symptoms. | Baseline to 8 weeks
  The number of participants with change in fatigue symptom on the Fatigue Severity Scale (FSS) score, total range score of 9-63, from baseline to week 8 in people with epilepsy (PWE)and moderate-to-severe insomnia with Go! To sleep (GTS) program compare to the number of participants with change in fatigue symptom on the Fatigue Severity Scale (FSS) score from baseline to week 8 in people with epilepsy (PWE) and moderate-to-severe insomnia without Go! To sleep (GTS) program
Secondary Aim 3 - To compare change in daytime sleepiness symptom on the Epworth Sleepiness Scale (ESS) from baseline to week 8 between Go! To sleep (GTS) and controls in people with epilepsy and moderate-to-severe insomnia symptoms. | Baseline to 8 weeks
  The number of participants with change in daytime sleepiness symptom on the Epworth Sleepiness Scale (ESS) score, total range score of 0-24, from baseline to week 8 in people with epilepsy (PWE)and moderate-to-severe insomnia with Go! To sleep (GTS) program compare to the number of participants with change in daytime sleepiness symptom on the Epworth Sleepiness Scale (ESS) score from baseline to week 8 in people with epilepsy (PWE) and moderate-to-severe insomnia without Go! To sleep (GTS) program
Secondary Aim 4 - To compare change in self-reported daily total sleep time (TST) from baseline to week 8 between Go! To sleep (GTS) and controls in people with epilepsy and moderate-to-severe insomnia symptoms. | Baseline to 8 weeks
  The number of participants with change in self-reported daily total sleep time (TST) (average of minutes of total sleep time in one week ) from baseline to week 8 in people with epilepsy (PWE)and moderate-to-severe insomnia with Go! To sleep (GTS) program compare to the number of participants with change self-reported daily total sleep time (TST) (average of minutes of total sleep time in one week ) from baseline to week 8 in people with epilepsy (PWE) and moderate-to-severe insomnia without Go! To sleep (GTS) program
Secondary Aim 5 - To compare change in depression symptom on the Patient Health Questionnaire-9 (PHQ-9) from baseline to week 8 between Go! To sleep (GTS) and controls in people with epilepsy and moderate-to-severe insomnia symptoms. | Baseline to 8 weeks
  The number of participants with change in depression symptom on the Patient Health Questionnaire-9 (PHQ-9) score, total range score of 0-27, from baseline to week 8 in people with epilepsy (PWE)and moderate-to-severe insomnia with Go! To sleep (GTS) program compare to the number of participants with depression symptom on the Patient Health Questionnaire-9 (PHQ-9) score from baseline to week 8 in people with epilepsy (PWE) and moderate-to-severe insomnia without Go! To sleep (GTS) program
Secondary Aim 6-To assess the relationship of change in sleep quality on the Pittsburgh Sleep Quality Inventory (PSQI) and adherence of Go! To sleep (GTS) program. | Baseline to 8 weeks
  The relationship between change in sleep quality on the Pittsburgh Sleep Quality Inventory (PSQI) score (total score range of 0-21), and the number of the day of participation and total number of lessons completed in Go! To sleep program in people with epilepsy (PWE) and moderate-to-severe insomnia with Go! To sleep (GTS) program.
Secondary Aim 7-To assess the relationship of change in fatigue symptom on the Fatigue Severity Scale (FSS) and adherence of Go! To sleep (GTS) program. | Baseline to 8 weeks
  The relationship between change in fatigue symptom on the Fatigue Severity Scale (FSS) score (total range score of 9-63), and the number of the day of participation and total number of lessons completed in Go! To sleep program in people with epilepsy (PWE) and moderate-to-severe insomnia with Go! To sleep (GTS) program.
Secondary Aim 8-To assess the relationship of change in daytime sleepiness symptom on the Epworth Sleepiness Scale (ESS) and adherence of Go! To sleep (GTS) program. | Baseline to 8 weeks
  The relationship between change in daytime sleepiness symptom on the Epworth Sleepiness Scale (ESS) score (total range score of 0-24), and the number of the day of participation and total number of lessons completed in Go! To sleep program in people with epilepsy (PWE) and moderate-to-severe insomnia with Go! To sleep (GTS) program.
Secondary Aim 9-To assess the relationship of change in self-reported daily total sleep time (TST) (average of minutes of total sleep time in one week) and adherence of Go! To sleep (GTS) program | Baseline to 8 weeks
  The relationship between change in self-reported daily total sleep time (TST) (average of minutes of total sleep time in one week) and the number of the day of participation and total number of lessons completed in Go! To sleep program in people with epilepsy (PWE) and moderate-to-severe insomnia with Go! To sleep (GTS) program.
Secondary Aim 10-To assess the relationship of change in depression symptom on the Patient Health Questionnaire-9 (PHQ-9) and adherence of Go! To sleep (GTS) program. | Baseline to 8 weeks
  The relationship between change in depression symptom on the Patient Health Questionnaire-9 (PHQ-9) score (total range score of 0-27) and the number of the day of participation and total number of lessons completed in Go! To sleep program in people with epilepsy (PWE) and moderate-to-severe insomnia with Go! To sleep (GTS) program.
Secondary Aim 11-To describe participant barrier to use the on-line Go! To sleep program by using Barrier to Computerized Cognitive Behavioral Therapy for Insomnia (CCBT-i) questionnaire | 8 weeks
  The people with epilepsy (PWE) and moderate-to-severe insomnia with Go! To sleep (GTS) program report barriers to use the on-line Go! To sleep (GTS) program by complete Barrier to Computerized Cognitive Behavioral Therapy for Insomnia (CCBT-i) questionnaire at week 8.
Secondary Aim 12-To compare change in sleep quality on the Pittsburgh Sleep Quality Inventory (PSQI) and mean daily seizure frequency from baseline to week 8 between GTS and controls in PWE and moderate-to-severe insomnia symptoms. | Baseline to 8 weeks
  The number of participants with change in sleep quality on the Pittsburgh Sleep Quality Inventory (PSQI)(total score range of 0-21),in both people with epilepsy (PWE)and moderate-to-severe insomnia with Go! To sleep (GTS) program and without Go! To sleep (GTS) program compare to change in total daily seizure frequency (amount of focal and generalized seizure per day) from baseline to week 8.
Secondary Aim 13-To compare change in fatigue symptom on the Fatigue Severity Scale (FSS) and mean daily seizure frequency from baseline to week 8 between GTS and controls in PWE and moderate-to-severe insomnia symptoms. | Baseline to 8 weeks
  The number of participants with change in fatigue symptom on the Fatigue Severity Scale (FSS) score (total range score of 9-63), in both people with epilepsy (PWE)and moderate-to-severe insomnia with Go! To sleep (GTS) program and without Go! To sleep (GTS) program compare to change in total daily seizure frequency (amount of focal and generalized seizure per day) from baseline to week 8.
Secondary Aim 14-To compare change in daytime sleepiness symptom on the Epworth Sleepiness Scale (ESS) and mean daily seizure frequency from baseline to week 8 between GTS and controls in PWE and moderate-to-severe insomnia symptoms. | Baseline to 8 weeks
  The number of participants with change in daytime sleepiness symptom on the Epworth Sleepiness Scale (ESS) score, total range score of 0-24, in both people with epilepsy (PWE)and moderate-to-severe insomnia with Go! To sleep (GTS) program and without Go! To sleep (GTS) program compare to change in total daily seizure frequency (amount of focal and generalized seizure per day) from baseline to week 8.
Secondary Aim 15-To compare change in self-reported daily total sleep time (TST) and mean daily seizure frequency from baseline to week 8 between GTS and controls in PWE and moderate-to-severe insomnia symptoms. | Baseline to 8 weeks
  The number of participants with change in self-reported daily total sleep time (TST) (average of minutes of total sleep time in one week ) in both people with epilepsy (PWE)and moderate-to-severe insomnia with Go! To sleep (GTS) program and without Go! To sleep (GTS) program compare to change in total daily seizure frequency (amount of focal and generalized seizure per day) from baseline to week 8.
Secondary Aim 16-To compare change in depression symptom on the Patient Health Questionnaire-9 (PHQ-9) and mean daily seizure frequency from baseline to week 8 between GTS and controls in PWE and moderate-to-severe insomnia symptoms. | Baseline to 8 weeks
  The number of participants with change in depression symptom on the Patient Health Questionnaire-9 (PHQ-9) score, total range score of 0-27, in both people with epilepsy (PWE)and moderate-to-severe insomnia with Go! To sleep (GTS) program and without Go! To sleep (GTS) program compare to change in total daily seizure frequency (amount of focal and generalized seizure per day) from baseline to week 8.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Foldvary-Schaefer, DO, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Main Campus, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided